CLINICAL TRIAL: NCT07399678
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study Assessing Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ALV-100 in Participants With Overweight or Obesity With or Without Type 2 Diabetes
Brief Title: Study of ALV-100 to Assess Safety, Tolerability, and PK/PD in Overweight/Obese Participants With or Without T2D
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alveus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALV-102-1
Record Dates: First submitted 2026-01-15; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Overweight or Obese Adults; Overweight or Obese, Type 2 Diabetes
Keywords: Overweight, Obese, Obesity, Type 2 Diabetes, Weight loss
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2; Weight Loss

STUDY DESIGN:
Intervention Model Description: In Part A, four treatment cohorts of participants with overweight or obesity will be administered varying dose escalation regimens of ALV-100. Each cohort will explore the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple doses of ALV-100. Each cohort will be comprised of 40 participants with 32 participants receiving active treatment and 8 participants receiving placebo in a 4:1 ratio.
  In Part B, a single cohort of participants with overweight or obesity, and T2D will be enrolled. This cohort will explore the safety (including glycemic safety), tolerability, pharmacokinetics, and pharmacodynamics of multiple doses of ALV-100. Fifteen (15) participants will receive active treatment, and 5 participants will receive placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part A - Cohort 1 (ALV-100) (Experimental): Participants with overweight or obesity without type 2 diabetes will receive ascending doses of ALV-100 by subcutaneous injection.
  Interventions: Drug: ALV-100
- Part A - Cohort 1 (Placebo) (Placebo Comparator): Participants with overweight or obesity without type 2 diabetes will receive placebo by subcutaneous injection.
  Interventions: Drug: Placebo
- Part A - Cohort 2 (ALV-100) (Experimental): Participants with overweight or obesity without type 2 diabetes will receive ascending doses of ALV-100 by subcutaneous injection.
  Interventions: Drug: ALV-100
- Part A - Cohort 2 (Placebo) (Placebo Comparator): Participants with overweight or obesity without type 2 diabetes will receive placebo by subcutaneous injection.
  Interventions: Drug: Placebo
- Part A - Cohort 3 (ALV-100) (Experimental): Participants with overweight or obesity without type 2 diabetes will receive ascending doses of ALV-100 by subcutaneous injection.
  Interventions: Drug: ALV-100
- Part A - Cohort 3 (Placebo) (Placebo Comparator): Participants with overweight or obesity without type 2 diabetes will receive placebo by subcutaneous injection.
  Interventions: Drug: Placebo
- Part A - Cohort 4 (ALV-100) (Experimental): Participants with overweight or obesity without type 2 diabetes will receive ascending doses of ALV-100 by subcutaneous injection.
  Interventions: Drug: ALV-100
- Part A - Cohort 4 (Placebo) (Placebo Comparator): Participants with overweight or obesity without type 2 diabetes will receive placebo by subcutaneous injection.
  Interventions: Drug: Placebo
- Part B - T2D Cohort (ALV-100) (Experimental): Participants with overweight or obesity with type 2 diabetes will receive ascending doses of ALV-100 by subcutaneous injection.
  Interventions: Drug: ALV-100
- Part B - T2D Cohort (Placebo) (Placebo Comparator): Participants with overweight or obesity with type 2 diabetes will receive placebo by subcutaneous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALV-100 — Participants will receive multiple ascending doses of ALV-100.
  Arms: Part A - Cohort 1 (ALV-100); Part A - Cohort 2 (ALV-100); Part A - Cohort 3 (ALV-100); Part A - Cohort 4 (ALV-100); Part B - T2D Cohort (ALV-100)
Drug: Placebo — Participants will receive placebo matching ALV-100, volume-matched to active dose.
  Arms: Part A - Cohort 1 (Placebo); Part A - Cohort 2 (Placebo); Part A - Cohort 3 (Placebo); Part A - Cohort 4 (Placebo); Part B - T2D Cohort (Placebo)

SUMMARY:
A Study of ALV-100 to Assess Safety, Tolerability, and PK/PD in Overweight/Obese Participants with or without Type 2 Diabetes

ELIGIBILITY:
Inclusion Criteria:

For Part A and B

* Adult male and female participants, aged 18 to 65 years, inclusive, at the time of signing the informed consent form
* Body mass index between 27.0 to 39.9 kg/m2 at Screening, both inclusive; overweight should be due to excess adipose tissue, as judged by the Investigator.
* Have a stable body weight (< 5.0 kg/11 lbs self-reported change) within 90 days prior to Screening
* Females must be surgically sterile (by means of bilateral salpingectomy, hysterectomy or bilateral oophorectomy) or be post-menopausal (defined as spontaneous cessation of menses for at least 1 year prior to Screening). Females who are post-menopausal and < 55 years must have a follicle-stimulating hormone level > 40 IU/L at Screening.
* Males with female partners of child-bearing potential must be willing to practice abstinence or must agree to use condom as contraception throughout the duration of the study. This criterion may be waived for male participants who have had a documented successful vasectomy > 6 months before signing the ICF.

For Part B only

* Diagnosis of Type 2 Diabetes for at least 180 days prior to Screening.
* Glycemic control managed by diet and exercise alone or by stable treatment with metformin and/or sodium-glucose cotransporter 2 inhibitors (SGLT-2i), with no dose changes within 3 months prior to Screening.
* Hemoglobin A1c (HbA1c) between 7.0 % and 9.0% (equivalent to 53-75 mmol/mol), both inclusive, at Screening.

Exclusion Criteria:

For Part A and B

* History or presence of any clinically relevant respiratory, metabolic (including dyslipidemia, however mild dyslipidemia, defined as screening total cholesterol below or equal to 302 mg/dL (7.8 mmol/L) and/or screening triglyceride below 300 mg/dL (3.39 mmol/L) is accepted), renal, hepatic, gastrointestinal, endocrinological conditions (except conditions associated with type 2 diabetes in Part B) at the discretion of the Investigator.
* Participants with a family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 or a personal history of nonfamilial medullary thyroid carcinoma.
* Current or history of chronic or acute pancreatitis.
* Obesity caused by known endocrinologic disorders (e.g., Cushing syndrome) or monogenetic or syndromic forms of obesity (for example, Melanocortin 4 Receptor deficiency or Prader Willi Syndrome).
* History of major depressive disorder or other severe psychiatric disorder (for example, schizophrenia, bipolar disorder, or anxiety disorder).
* Lifetime history of a suicide attempt or of any suicidal behavior by endorsement of (answered yes to) any of the items in the suicidal behavior section on the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening.
* Systolic blood pressure ≥ 140 mm Hg or diastolic blood pressure ≥ 90 mm Hg at Screening.
* History of or current cardiovascular disease, including but not limited to stable and unstable angina, myocardial infarction, congestive heart failure, transient ischemic attack, stroke, clinically significant arrhythmias and conduction disorders or venous thromboembolism.

Part A only

• History or clinical evidence of Type 1 or Type 2 diabetes mellitus, including HbA1c ≥ 6.5% and/or a fasting plasma glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L) at Screening (female participants with a history of gestational diabetes are allowed).

Part B only

* Fasting plasma glucose (FPG) > 270 mg/dL (15.0 mmol/L) at Screening.
* Proliferative retinopathy or maculopathy as judged by the investigator based on a recent (within1.5 years from Screening) ophthalmologic examination.
* Severe neuropathy as judged by the investigator.
* Advanced nephropathy (defined as albuminuria ≥ 300 mg/g).
* History of severe hypoglycemia or hypoglycemic unawareness as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | From First Dose to Week 52
  Incidence of treatment emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of intact ALV-100 and total ALV-100 - Cmax, MD | From First Dose to Week 52
  Maximum observed serum concentration after multiple doses (MD) (Cmax, MD)
Pharmacokinetics (PK) of intact ALV-100 and total ALV-100 - AUC(0-τ), MD | From First Dose to Week 52
  Area under the serum concentration-time curve from time zero to the last quantifiable concentration (AUC(0-τ), MD)
Pharmacodynamic (PD) impact on body weight | Baseline, Week 32 and Week 52
  Change from baseline in body weight
Pharmacodynamic (PD) impact on body weight percentage | Baseline, Week 32 and Week 52
  Change from baseline in body weight percentage
Immunogenicity | From Baseline to Week 52
  Incidence of Anti-ALV-100 drug antibodies, including assessments of cross-reactivity and neutralizing antibodies.
Relationship between ALV-100 serum concentration and QTc interval changes (Part A Only) | From First Dose to Week 52
  Measurement of change in individual specific heart rate corrected QT interval (QTcI) and Fridericia heart rate corrected QT interval (QTcF) on 12-lead ECG.
Paracetamol (acetaminophen) absorption test (PAT) (Part A Only) | From First Dose to Week 52
  Measurement of acetaminophen PK parameters to evaluate the effect of ALV-100 on the gastric emptying rate.
Pharmacodynamic (PD) impact of ALV-100 on antidiabetic medication (Part B Only) | From Baseline to Week 32
  Change in use of concomitant glucose-lowering medication
Pharmacodynamic (PD) impact of ALV-100 on glycemic parameters (Part B Only) | Week 32 and Week 52
  Measuring the number of participants achieving target Hemoglobin A1c values
Hypoglycemic Safety (Part B Only) | From Baseline to Week 52
  Measured by the incidence of symptomatic hypoglycemia, documented symptomatic hypoglycemia and severe hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Karen Tornøe, MD, PhD, Study Director — Alveus Therapeutics
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No